CLINICAL TRIAL: NCT01001910
Title: Phase II Trial of Combination Pemetrexed (Alimta) and Carboplatin (Paraplatin) in Platinum Sensitive Recurrent Ovarian, Primary Peritoneal, and Fallopian Tube Carcinoma
Brief Title: Pemetrexed and Carboplatin in Treating Patients With Recurrent Ovarian, Primary Peritoneal, or Fallopian Tube Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-04-097; NCI-2013-01208 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 08-015; 08-04-097 (Other: Albert Einstein College of Medicine); P30CA013330 (NIH)
Record Dates: First submitted 2009-10-26; First posted 2009-10-27 (Estimated); Results first posted 2021-10-20 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Carboplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (pemetrexed disodium, carboplatin) (Experimental): Patients receive pemetrexed disodium IV over 8-15 minutes and carboplatin IV over 30-60 minutes on day 1. Treatment repeats every 21 days for at least 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Other: Laboratory Biomarker Analysis; Drug: Pemetrexed Disodium

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplat; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Pemetrexed Disodium — Given IV
  Other Names: Alimta; LY231514; N-[4-[2-(2-Amino-4,7-dihydro-4-oxo-1H-pyrrolo[2,3-d]pyrimidin-5-yl)ethyl]benzoyl]-L-glutamic Acid Disodium Salt

SUMMARY:
This phase II trial studies how well pemetrexed disodium and carboplatin work in treating patients with recurrent ovarian, primary peritoneal, or fallopian tube cancer. Drugs used in chemotherapy, such as pemetrexed disodium and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the response rate of combination pemetrexed (pemetrexed disodium) (Alimta) and carboplatin (Paraplatin) in recurrent ovarian, primary peritoneal, and fallopian tube carcinoma.

SECONDARY OBJECTIVES:

I. To evaluate the progression free interval, overall survival, and adverse effects among patients receiving this drug combination.

OUTLINE:

Patients receive pemetrexed disodium intravenously (IV) over 8-15 minutes and carboplatin IV over 30-60 minutes on day 1. Treatment repeats every 21 days for at least 6 courses in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histopathologically confirmed diagnosis of epithelial ovarian, primary peritoneal, or fallopian tube carcinoma
* Patients must have received at least 1 prior platinum and taxane based chemotherapy regimen; patients may have failed no more than 2 prior chemotherapy regimens
* Patients must have "platinum sensitive" disease, which will be defined as those patients with relapsed disease who had an initial complete remission, and relapsed more than 6 months after completion of initial platinum based chemotherapy
* Recurrent disease must be confirmed by:

  * Bidimensionally measurable disease which can be measured by physical examination or by means of medical imaging techniques (measurable disease)

    * Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest dimension to be recorded); each lesion must be >= 2.0 cm when measured by conventional techniques, including palpation, x-ray, computed tomography (CT), and magnetic resonance imaging (MRI), or >= 1.0 cm when measured by spiral CT; all measurable lesions up to a maximum of 5 lesions per organ and 10 lesions in total representative of all involved organs should be identified as target lesions and will be recorded and measured at baseline; all baseline evaluations of disease status should be performed as close as possible to the start of treatment and never more than 4 weeks before the beginning of treatment
    * Target lesions should be selected on the basis of their size (lesions with the longest dimension, LD) and their suitability for accurate repetitive measurements by one consistent method of assessment (either clinically or by imaging techniques); a sum of LD for all target lesions will be calculated and reported as the baseline sum LD; the baseline sum LD will be used as reference to further characterize the objective tumor response of the measurable dimension of the disease; all other lesions (or sites of disease) should be identified as non-target lesions and should also be recorded at baseline OR
  * Two confirmed serum cancer antigen-125 (CA-125) levels greater than or equal to 70 u/ml (or 2 x upper limit of normal) separated by 1 week and obtained within 4 weeks prior to entry to the study (evaluable disease)
* Patients must not have had other myelosuppressive therapy within four weeks of initiating pemetrexed/ carboplatin therapy
* Patients must have recovered from effects of recent surgery
* Patients must have a Gynecologic Oncology Group (GOG) performance status of 0, 1, or 2
* White blood cell (WBC) greater than or equal to 3,000/ul
* Platelet count greater or equal to 100,000/ul
* Neutrophil count greater or equal to 1,500/ul
* Creatinine clearance >= 45 ml/min (estimated creatinine clearance by Cockcroft-Gault equation acceptable)
* Total bilirubin =< to 1.5 mg/dL
* Serum glutamic oxaloacetic transaminase (SGOT) and serum glutamate pyruvate transaminase (SGPT) =< three times the upper normal institutional limits; if patient has known hepatic metastases, patients may be enrolled if liver function test is =< five times the upper normal institutional limits
* Alkaline phosphatase =< three times the upper normal institutional limits; if patient has known hepatic metastases, patients may be enrolled if liver function test is =< five times the upper normal institutional limits
* Patient must have signed informed consent
* Patients must be willing to take the dexamethasone, folic acid and vitamin B12 supplementation as indicated in the protocol to reduce adverse drug toxicity
* Patients must be willing to interrupt aspirin and other nonsteroidal anti-inflammatory drugs (NSAID) intake for 2 days before, day of, and 2 days after each chemotherapy treatment; low dose 80 mg aspirin and cyclooxygenase-2 (Cox-2) inhibitors are excluded from this restriction; if concomitant administration of an NSAID is necessary, patients should be monitored closely
* Patients must have a life expectancy of greater than 12 weeks
* Patients may not have concurrent or previous invasive malignancies, with the exception of non-melanoma skin cancer or no evidence of recurrence of previous malignancy within the last 5 years
* Patients must have a current exam, blood work and any clinically indicated imaging studies within 4 weeks prior to study enrollment
* Baseline folate and homocysteine blood levels
* The ability to interrupt NSAIDS 2 days before (5 days for long-acting NSAIDs), the day of, and 2 days following administration of Alimta
* The ability to take folic acid, vitamin B12, and dexamethasone according to protocol

Exclusion Criteria:

* Patients who have had more than two prior chemotherapeutic regimens
* Patients who have had prior treatment with pemetrexed
* Patients with a GOG performance status of 3 or 4
* Patients with >= grade 2 neuropathy
* Patients who have received external beam whole pelvic or whole abdominal radiation treatment (>= 4500 centigray [cGy]) which would limit vascular capacity and reduce adequate drug delivery
* Patients with evidence of recurrence from another malignancy within the previous five years
* Patients with a concomitant malignancy other than squamous cell skin cancer
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients who have received an investigational drug within the last 30 days that has not received regulatory approval
* Presence of third space fluid which cannot be controlled by drainage; for patients who develop or have baseline clinically significant pleural or peritoneal effusions (on the basis of symptoms or clinical examination) before or during initiation of Alimta therapy, consideration should be given to draining the effusion prior to dosing; however, if, in the investigator's opinion, the effusion represents progression of disease, the patient should be discontinued from study therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-07; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Kuo, Principal Investigator — Albert Einstein College of Medicine
Locations (3):
- United States (3):
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Albert Einstein College of Medicine, The Bronx, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The sample size calculation was based on the primary endpoint of ORR. According to the Simon 2 stage design, the maximum trial size was set at 46 evaluable patients and stopping rules were based on the error probability limits of α=0.05 and β=0.1. If < 8 responses were observed among the initial 22 patients, the study would be terminated.
Period: Overall Study
Arm/Group | Treatment (Pemetrexed Disodium, Carboplatin)
Started | 28 (We screened and started 28 patients in the study. However only 22 patients were evaluable for outcome, because 6 patients did not receive adequate number of cycles of treatment for analysis. While we could not evaluate these 6 patients for their outcome, their treatment-cycles were included in the safe analysis.)
Completed | 22 (6 patients did not receive 3 cycles required for evaluation of response as per protocol s7.1.1)
Not Completed | 6
Not completed — Did not meet protocol defined eligibility s7.1.1 for primary outcome | 6

BASELINE CHARACTERISTICS:
Population: This is a open-labeled, phase II trial evaluating the combination of intravenous pemetrexed and carboplatin in patients with confirmed recurrent epithelial ovarian, primary peritoneal, or fallopian tube carcinoma. There is no comparison group.
Arm/Group | Treatment (Pemetrexed Disodium, Carboplatin)
Number analyzed (Participants) | 28
Age, Continuous [Median (Full Range); unit: years] | 64 [46 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 21
  Race: African American | 1
  Race: Hispanic | 3
  Race: Asian | 3
Site of Disease [Count of Participants; unit: Participants]
  Ovary | 23
  Primary Peritoneal | 4
  Fallopian Tube | 1
FIGO Stage at Diagnosis [Count of Participants; unit: Participants] — The stage reported here for the patients enrolled was the stage at their initial diagnosis. Surgical staging was performed primarily for the patients. Patients with Stage I disease had tumor spread that was confined to the pelvis. Patients with Stage II disease had tumor spread to organs/tissues surrounding the pelvis. Patients with Stage III had tumor spread to distant nodes or tissue within the pelvis. Patients with Stage IV disease had tumor spread to the upper abdomen, retroperitoneum, or other distant organs including lung and liver.
  Participants
    Stages I/II | 3
    Stages III/IV | 25

OUTCOME MEASURES:

1. Primary Outcome: Overall Objective Response Rate (ORR) Based on Response Evaluation Criteria in Solid Tumors and by Rustin's Criteria (RECIST)
Description: The primary endpoint is overall response rate defined by proportion of patients achieving complete response, partial response based on RECIST V1.1 or Rustin's criteria as appropriate.
  Based on RECIST V1.1 for targeting lesions from CT scan: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions; Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study; Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD; Overall response CR + PR.
  Based on Rustin's criteria, a response to ca125 has occurred if there is at least a 50% reduction in ca125 level from a pretreatment sample. The response must be confirmed and maintained for at least 28 days.
Time Frame: 4.5 years
Population: Intent to Treat Patients were included for primary endpoint analysis of ORR if they completed 3 cycles of therapy. Response was categorized as complete response (CR), partial response (PR), stable disease (SD) or progressive disease (PD) by RECIST criteria. All patients had
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pemetrexed Disodium, Carboplatin)
Number analyzed (Participants) | 22
Participants
  Complete response | 4
  Partial response | 5
  Stable disease | 9
  Progressive disease | 4

2. Secondary Outcome: Incidence of Toxicities
Description: Secondary outcome included detailed measurement of adverse events from treatment assessed according to National Cancer Institute (NCI) Common Toxicity Criteria (CTC) version 3.0.
Time Frame: 4.5 years
Population: The patients that received pemetrexed disodium with carboplatin treatment were evaluated for an grade, grade 3, and grade 4 toxicities for adverse event confirmations.
Measure: Number; unit: Frequency of event
Arm/Group | Treatment (Pemetrexed Disodium, Carboplatin)
Number analyzed (Participants) | 22
Frequency of event
  Hematologic AE Any Grade | 240
  Non-Hematologic AE Any Grade | 60

3. Secondary Outcome: Overall Survival (OS)
Description: Kaplan-Meier method will be used t analyze the time-to-event data including overall survival (OS) and progression-free survival (PFS)
Time Frame: First day of treatment on protocol to the date of death, or for living patients the last date of contact, assessed up to 4.5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Pemetrexed Disodium, Carboplatin)
Number analyzed (Participants) | 22
months
  PFS | 6.8 [5.1 to 8.7]
  OS | 50.3 [17.1 to 55.1]

4. Secondary Outcome: Progression-free Interval
Description: Kaplan-Meier curve will be used to examine all the time-to-event data points in analyzing progression free interval.
Time Frame: Time from the first day of treatment to the day that progression is first noted, assessed up to 4.5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Pemetrexed Disodium, Carboplatin)
Number analyzed (Participants) | 22
months | 6.8 [5.1 to 8.7]

ADVERSE EVENTS:
Time Frame: The median exposure to combination pemetrexed and carboplatin therapy was 18.9 weeks (range: 3-37.9 weeks). The safety population included all patients who received one cycle of chemotherapy and was included in the analysis of safety data.
Description: Adverse events were graded on a scale of 1 to 4, for unfavorable medical occurrences in a participant whether or not considered related to the participant's participation in the research. The types of toxicities evaluated consisted of "hematologic" versus "non-hematologic." Treatment related deaths were recorded separately from all-cause mortality cases. Frequency of adverse events are calculated based on the total number of events divided by the total number of chemotherapy cycles given.
Arm/Group | Treatment (Pemetrexed Disodium, Carboplatin)
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 11/22
Other Adverse Events (participants affected / at risk) | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pemetrexed Disodium, Carboplatin) (N=22)
Hematologic (Blood and lymphatic system disorders) | 8 (71) — Neutropenia or Thrombocytopenia or Anemia
Non-Hematologic (General disorders) | 3 (15) — Elevated LFTs or Abdominal pain or Hypomagnesemia or Hyperglycemia or Hypersensitivity or Chest pain or Temporal parietal hemotoma or Bell's palsy

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes